CLINICAL TRIAL: NCT05394701
Title: Comparing the Pharmacological Profile of Enteric Coated and Non-Enteric Coated Capsules Containing Omega 3 Fatty Acids
Brief Title: Comparing the Pharmacological Profile of Formulations Containing Omega 3 Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Factors Group of Nutritional Companies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10-002
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pharmacokinetics
Keywords: Bioavailability; Pharmacokinetics; Omega-3 fatty acids; Fish Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RxOmega-3 soft gels (Enteric) (Experimental): Each participant receives their treatment of RxOmega-3 soft gel (Enteric) capsules at a total dose of 1260 mg Omega-3 Fatty Acids. Treatments are consumed with a glass of water (approx. 200 mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours.
  Participants are asked to arrive after an overnight fast (at least 9hrs). Each participant acts as their own control; there is no separate control group. A washout period of at least 14 days between each treatment will be used.
  Adverse events are recorded throughout the study by direct questioning.
  Interventions: Dietary Supplement: RxOmega-3 soft gels (Enteric)
- Omega-3 Complete soft gels (Non-Enteric) (Experimental): Each participant receives their treatment of Omega-3 Complete soft gel (Non-Enteric) capsules at a total dose of 1260 mg Omega-3 Fatty Acids. Treatments are consumed with a glass of water (approx. 200 mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours.
  Participants are asked to arrive after an overnight fast (at least 9hrs). Each participant acts as their own control; there is no separate control group. A washout period of at least 14 days between each treatment will be used.
  Adverse events are recorded throughout the study by direct questioning.
  Interventions: Dietary Supplement: Omega-3 Complete soft gels (Non-Enteric)
- Omega-3 LipoMicel® soft gels (Experimental): Each participant receives their treatment of Omega-3 LipoMicel® soft gel capsules at a total dose of 1260 mg Omega-3 Fatty Acids. Treatments are consumed with a glass of water (approx. 200 mL), followed by a standardized breakfast (diet-controlled condition). Capillary whole blood samples are collected at time points 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours.
  Participants are asked to arrive after an overnight fast (at least 9hrs). Each participant acts as their own control; there is no separate control group. A washout period of at least 14 days between each treatment will be used.
  Adverse events are recorded throughout the study by direct questioning.
  Interventions: Dietary Supplement: Omega-3 LipoMicel® soft gels

INTERVENTIONS:
Dietary Supplement: Omega-3 LipoMicel® soft gels — A maximum single dose of 1260 mg Omega-3 Fatty Acids: Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA)
  Arms: Omega-3 LipoMicel® soft gels
Dietary Supplement: RxOmega-3 soft gels (Enteric) — A maximum single dose of 1260 mg Omega-3 Fatty Acids: Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA)
  Arms: RxOmega-3 soft gels (Enteric)
Dietary Supplement: Omega-3 Complete soft gels (Non-Enteric) — A maximum single dose of 1260 mg Omega-3 Fatty Acids: Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA)
  Arms: Omega-3 Complete soft gels (Non-Enteric)

SUMMARY:
The primary objective of this study is to investigate the uptake/gastrointestinal absorption of fatty acids in healthy adult volunteers by using enteric coated and non-enteric coated soft capsules containing omega 3 fatty acids. Pharmacokinetic parameters such as AUC and Cmax, as well as any adverse events are recorded.

As secondary objective, the short-term effects of Omega-3 supplementation on blood lipid parameters in healthy volunteers are evaluated using a Cholestech LDX analyzer to measure cholesterol and related lipids.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* healthy, good physical condition

Exclusion Criteria:

* Pregnancy or breast-feeding
* Gastrointestinal conditions
* Acute or chronic liver disease
* Acute or chronic kidney disease
* Acute or chronic cardiovascular disease
* Allergy or Intolerance to gluten
* Allergy or Intolerance to fish or shellfish
* Use of medications (e.g., anticoagulants/ blood thinners such as warfarin; blood lipid-lowering agents such as statins)
* Use of Fish oil supplements
* Use of any form of nicotine or tobacco
* Alcohol and substance abuse history
* Participation in another investigational study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
AUC: the area under the concentration-time curve | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested omega-3 fatty acids in enteric coated soft gel capsules in healthy adult volunteers and compare the Area under the plasma concentration versus time curve (AUC) with that of non-enteric coated soft capsules containing omega 3 fatty acids.
Cmax: maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested omega-3 fatty acids in enteric coated soft gel capsules in healthy adult volunteers and compare the Peak Plasma Concentration (Cmax) with that of non-enteric coated soft capsules containing omega 3 fatty acids.
Tmax: the time point of maximum plasma concentration | 0 (baseline; pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24 hours (post-dose)
  To determine the gastrointestinal absorption of orally ingested omega-3 fatty acids in enteric coated soft gel capsules in healthy adult volunteers and compare the time point of maximum plasma concentration (Tmax) with that of non-enteric coated soft capsules containing omega 3 fatty acids.

SECONDARY OUTCOMES:
Effects on blood lipid parameters | 0 (Baseline; pre-dose), 3, 6, 12, 24, 48, 72, 96, 120 hours post-dose
  To evaluate the short-term effects of orally ingested omega-3 fatty acids on cholesterol levels in healthy volunteers by using a Cholestech LDX analyzer.
Changes in blood lipid concentrations | 0 (Baseline; pre-dose), 3, 6, 12, 24, 48, 72, 96, 120 hours post-dose
  To evaluate changes in blood lipid concentrations of orally ingested omega-3 fatty acids in healthy volunteers by using a Cholestech LDX analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Solnier, PhD, Principal Investigator — Isura
Locations (1):
- ISURA, Burnaby, British Columbia, Canada